CLINICAL TRIAL: NCT04453878
Title: Using Ultrasound-guide Corrected Glenohumeral Internal Rotation Deficit as a Risk Factor to Predict Shoulder Injuries in Baseball Players
Brief Title: Ultrasound-guide Corrected Glenohumeral Internal Rotation Deficit
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202005109RINB
Record Dates: First submitted 2020-06-22; First posted 2020-07-01 (Actual); Last update posted 2023-10-18 (Actual); Status verified 2023-10

CONDITIONS: Glenohumeral Internal Rotation Deficit
Keywords: shoulder injury,ultrasound
MeSH Terms: conditions — Shoulder Injuries

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Background:

Glenohumeral internal rotation deficit (GIRD) is believed to be one of the risk factors contributing to shoulder injuries. In addition, athletes with GIRD of greater than 20° appear to be at a greater risk for the shoulder injuries and surgery. Recently, GIRD can be divided in anatomical GIRD and pathological GIRD (pGIRD). The dominant arm of the athletes with pGIRD have not only humeral retrotorsion (HR) but also stiffer posterior capsule. The soft-tissue effect is believed to be the key point in pathological cascade of throwers. Therefore, the previous studies use gross GIRD as a risk factor may be modified by ultrasound-guide corrected GIRD.

Objective:

There are 4 objectives for the present study: (1) to investigate the Receiver operating characteristic (ROC) curves of the gross GIRD; (2) to investigate the ROC curves of the ultrasound-guide corrected GIRD; (3) to compare the area under curve (AUC) of the two methods; (4) to compare the gross GIRD and the ultrasound-guide corrected GIRD in baseball players.

Design:

Baseball players who have played baseball for at least 1 year and still active in training or competition will be recruited in this study. Participant characteristics will be collected by the main assessor, including age, gender, height, weight, dominant arm, practice time, years of playing baseball. Performance/function will be assessed via a Kerlan-Jobe Orthopaedic Clinic shoulder and elbow (KJOC) self-report questionnaire. The shoulder rotation ROM, ultrasound examination including ultrasound-corrected GIRD and posterior capsular thickness and posterior shoulder tightness will also be measured. we will follow subjects for a season. Once the injury occurs, deterioration or at the end of the season, we will collect the data again.

Main outcome measures:

The shoulder rotation ROM, ultrasound examination and posterior shoulder tightness are main outcomes of the study.

ELIGIBILITY:
Inclusion criteria:

1. Age range from 12 to 40 years old.
2. Playing baseball for at least 1 year.
3. Still active in training or competition.
4. The frequency of training or game should be at least 3 times per week, 3 hours per time.

Exclusion criteria:

1. Subjects with shoulder pain onset due to trauma.
2. A history of shoulder fractures or dislocation.
3. Cervical radiculopathy.
4. Degenerative joint disease of the shoulder.
5. Surgical interventions on the shoulder.
6. Inflammatory arthropathy.

Ages: 12 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: A baseball team usually consists of 30 to 40 players. Therefore, we will recruit 3 or 4 local baseball teams in Taipei and New Taipei city. Based on the consideration of schedule between baseball teams and our research team, We will collect 7 subjects per day and the recruitment time will last for about a month.
Sampling Method: Probability Sample
Enrollment: 106 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-10-27 (Actual); Study Completion 2021-10-27 (Actual)

PRIMARY OUTCOMES:
alteration of ultrasound-guide corrected GIRD | through study completion, an average of 1 year
  The participants will be told to supine with 90° of shoulder abduction and elbow flexion. The main assessor places the transducer on the subject's anterior shoulder, perpendicular to the long axis of the humerus in the frontal plane. Then, the humerus will be manually rotated by the assessor for the bicipital groove being centered on the ultrasound image. The ultrasound is then positioned, aided by use of a grid on the ultrasound display. Thus, a line connecting the greater and lesser tubercles can be parallel to the horizontal plane. Last, the second assessor places a digital inclinometer on the ulnar side of the forearm to record the forearm inclination angle, defining the amount of humeral retroversion. This measurement will be repeated 3 times bilaterally and the average will be used for data analysis. The equation of ultrasound-guide corrected GIRD will be gross GIRD minus difference of humeral retroversion between dominant and non-dominant arm.
alteration of posterior capsular thickness | through study completion, an average of 1 year
  The subject will be positioned upright in a chair with the arm at the side and forearm resting on the thigh. The examiner positions a transducer on the posterior shoulder, visualizing the glenoid labrum, humeral head, rotator cuff, and posterior capsule, defined as the tissue immediately lateral to the tip of the labrum between the humeral head and rotator cuff. When the capsule is identified, the image is paused, and the capsule thickness will be measured by built-in caliper. The imaging procedure will be repeated 3 times, and an average thickness will be determined. This measurement will be taken bilaterally for all subjects.

SECONDARY OUTCOMES:
change of shoulder rotation ROM | through study completion, an average of 1 year
  Subjects will be placed in supine with the shoulder at 90° of abduction and elbow at 90° of flexion. The main assessor stabilizes the scapula then passively rotating the forearm internally or externally until end feel is reached. Another assessor places a digital inclinometer on the dorsal or the ventral side of the forearm to record the data. Each measurement will be performed 3 times both in the dominant and non-dominant arm, and the average data on the dominant and non-dominant sides will be used for analysis. The total rotation ROM will be the sum of the IR and external rotation.
Injury assessment and classification | up to 24 weeks
  The process will be modified according to the previous studies. The players will be prospectively tracked for overuse shoulder injuries throughout the season. For the asymptomatic subjects, any complaint of shoulder problems reported by coach, parents or player will be evaluated by a physical therapist to verify the injury. Moreover, less than 70 KJOC score will be recognized as injury. Injury that does not occur during participation or unrelated to baseball will be excluded. For the symptomatic subject, if he feels exacerbation of the symptom, he will be told to report KJOC score again. Once the decreased score is over 30, the subject will be recognized as injury.
change of posterior shoulder tightness | through study completion, an average of 1 year
  To begin the test, the tester grasps the subject's extremity distal to the epicondyles of the elbow in supine position. The humerus will be passively moved into the starting position of 90˚ of flexion (if not possible, maximal flexion position) and 0˚ of adduction with neutral rotation for assessment of posterior shoulder tightness. At this point, the scapula will be palpated at the lateral border and stabilized with the hand. While the scapula is stabilized, the humerus is then passively moved into a cross-chest adduction with neutral rotation. The humerus is moved until the movement cease (firm end-feel), indicating the end of shoulder tissue flexibility. The recorder places the digital inclinometer parallel to the humerus next to the medial epicondyle. The measured angle indicates the amount of flexibility of the posterior shoulder tissues. A greater angle indicates more flexibility of the shoulder tissue.
change of Kerlan-Jobe Orthopaedic Clinic Shoulder and Elbow score (KJOC) | through study completion, an average of 1 year
  The KJOC is the most common questionnaire for overhead athletes which has been conducted in several studies. Recently, Major League Baseball (MLB) organization also adopts this evaluation tool as the standard for the recovery of injuries in MLB players. The questionnaire is commonly used to assess shoulder function and performance. It is valid, reliable in its pilot form, and responsive in the tested population of adult overhead athletes. KJOC questionnaire range from 0 to 100 and the lower score represents limited function.
days in the disable list | through study completion, an average of 1 year
  The number of days that players cannot participate in the training or game due to injury will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Jing-Lan Yang, MAMS, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

REFERENCES:
- [Background] 1. Olsen SJ, 2nd, Fleisig GS, Dun S, Loftice J, Andrews JR. Risk factors for shoulder and elbow injuries in adolescent baseball pitchers. The American journal of sports medicine 2006;34:905-12. 2. Makhni EC, Morrow ZS, Luchetti TJ, Mishra-Kalyani PS, Gualtieri AP, Lee RW, et al. Arm pain in youth baseball players: a survey of healthy players. The American journal of sports medicine 2015;43:41-6. 3. Saper MG, Pierpoint LA, Liu W, Comstock RD, Polousky JD, Andrews JR. Epidemiology of Shoulder and Elbow Injuries Among United States High School Baseball Players: School Years 2005-2006 Through 2014-2015. The American journal of sports medicine 2018;46:37-43. 4. Dick R, Sauers EL, Agel J, Keuter G, Marshall SW, McCarty K, et al. Descriptive epidemiology of collegiate men's baseball injuries: National Collegiate Athletic Association Injury Surveillance System, 1988-1989 through 2003-2004. J Athl Train 2007;42:183-93. 5. Conte S, Camp CL, Dines JS. Injury Trends in Major League Baseball Over 18 Seasons: 1998-2015. Am J Orthop (Belle Mead NJ) 2016;45:116-23. 6. Lin DJ, Wong TT, Kazam JK. Shoulder Injuries in the Overhead-Throwing Athlete: Epidemiology, Mechanisms of Injury, and Imaging Findings. Radiology 2018;286:370-87. 7. Tyler TF, Nicholas SJ, Lee SJ, Mullaney M, McHugh MP. Correction of posterior shoulder tightness is associated with symptom resolution in patients with internal impingement. The American journal of sports medicine 2010;38:114-9. 8. Wilk KE, Macrina LC, Fleisig GS, Porterfield R, Simpson CD, 2nd, Harker P, et al. Correlation of glenohumeral internal rotation deficit and total rotational motion to shoulder injuries in professional baseball pitchers. The American journal of sports medicine 2011;39:329-35. 9. Harryman DT, 2nd, Sidles JA, Clark JM, McQuade KJ, Gibb TD, Matsen FA, 3rd. Translation of the humeral head on the glenoid with passive glenohumeral motion. The Journal of bone and joint surgery American volume 1990;72:1334-43. 10. Ludewig PM, Cook TM. Alterations in shoulder kinematics and associated muscle activity in people with symptoms of shoulder impingement. Physical therapy 2000;80:276-91. 11. Lin JJ, Hanten WP, Olson SL, Roddey TS, Soto-quijano DA, Lim HK, et al. Functional activity characteristics of individuals with shoulder dysfunctions. Journal of electromyography and kinesiology : official journal of the International Society of Electrophysiological Kinesiology 2005;15:576-86. 12. Itoi E, Motzkin NE, Morrey BF, An KN. Scapular inclination and inferior stability of the shoulder. Journal of shoulder and elbow surgery 1992;1:131-9. 13. Paley KJ, Jobe FW, Pink MM, Kvitne RS, ElAttrache NS. Arthroscopic findings in the overhand throwing athlete: evidence for posterior internal impingement of the rotator cuff. Arthroscopy : the journal of arthroscopic & related surgery : official publication of the Arthroscopy Association of North America and the International Arthroscopy Association 2000;16:35-40. 14. Warner JJ, Micheli LJ, Arslanian LE, Kennedy J, Kennedy R. Scapulothoracic motion in normal shoulders and shoulders with glenohumeral instability and impingement syndrome. A study using Moire topographic analysis. Clinical orthopaedics and related research 1992:191-9. 15. Weiser WM, Lee TQ, McMaster WC, McMahon PJ. Effects of simulated scapular protraction on anterior glenohumeral stability. The American journal of sports medicine 1999;27:801-5. 16. Kolber MJ, Hanney WJ. The reliability and concurrent validity of shoulder mobility measurements using a digital inclinometer and goniometer: a technical report. International journal of sports physical therapy 2012;7:306-13.